CLINICAL TRIAL: NCT00027599
Title: A Phase II Study Of Prostatic Acid Phosphatase-Pulsed Dendritic Cells (Provenge) In Combination With Bevacizumab In Patients With Serologic Progression Of Prostate Cancer After Definitive Local Therapy
Brief Title: APC8015 and Bevacizumab in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02427; UCSF-0155-01; NCI-2617; UCSF-01554; CDR0000069047 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-12-07; First posted 2003-05-07 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; sipuleucel-T

ARMS (1):
- Arm I (Experimental): Autologous dendritic cells (DCs) are harvested and pulsed with prostatic acid phosphatase-sargramostim fusion protein to produce APC8015 (Provenge). Patients receive APC8015 IV over 30 minutes and bevacizumab IV over 30-60 minutes on day 1. Treatment repeats every 14 days for 3 courses. Patients continue to receive bevacizumab alone every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Biological: prostatic acid phosphatase-sargramostim fusion protein; Biological: sipuleucel-T; Biological: therapeutic autologous dendritic cells; Procedure: in vitro-treated peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: bevacizumab
Biological: prostatic acid phosphatase-sargramostim fusion protein
Biological: sipuleucel-T
Biological: therapeutic autologous dendritic cells
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
Phase II trial to study the effectiveness of APC8015 combined with bevacizumab in treating patients who have undergone radiation therapy and/or surgery and who have progressive prostate cancer. Biological therapies such as APC8015 use different ways to stimulate the immune system and stop cancer cells from growing. Monoclonal antibodies such as bevacizumab can locate tumor cells and kill them without harming normal cells. Combining monoclonal antibody therapy with biological therapy may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of APC8015 (Provenge) and bevacizumab, in terms of decline in prostate-specific antigen (PSA) value and effect on PSA doubling time, in patients with progressive prostate cancer.

II. Determine any immune response in patients treated with this regimen. III. Determine the safety of this regimen in these patients.

OUTLINE:

Autologous dendritic cells (DCs) are harvested and pulsed with prostatic acid phosphatase-sargramostim fusion protein to produce APC8015 (Provenge). Patients receive APC8015 IV over 30 minutes and bevacizumab IV over 30-60 minutes on day 1. Treatment repeats every 14 days for 3 courses. Patients continue to receive bevacizumab alone every 14 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Any T, any N, M0
* Received prior therapy comprising one of the following regimens for primary prostate cancer:

  * External beam radiotherapy
  * Brachytherapy with or without pelvic external beam radiotherapy
  * Cryosurgery
  * Radical prostatectomy with or without adjuvant or salvage radiotherapy

    * Adjuvant or salvage radiotherapy after radical prostatectomy is allowed provided the following criteria is met:

      * PSA was never greater than 6.0 ng/mL
      * At least 3 months since androgen deprivation
* Elevated PSA (0.4-6.0 ng/mL) that has increased on 2 measurements taken at least 2 weeks apart
* No history of or radiological evidence of current CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, or brain metastases)

PATIENT CHARACTERISTICS:

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 months

Hematopoietic:

* WBC greater than 2,500/mm^3
* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* No prior bleeding disorder

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 2 times ULN
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 2 times ULN
* BUN no greater than 2 times ULN

Cardiovascular:

* No clinically significant cardiovascular disease
* No New York Heart Association grade II-IV heart disease (symptomatic congestive heart failure)
* No unstable angina pectoris
* No serious cardiac arrhythmia requiring medication
* No uncontrolled hypertension
* No prior myocardial infarction
* No grade II or greater peripheral vascular disease within the past year
* No prior deep vein thrombosis

Other:

* Fertile patients must use effective contraception
* HIV and HTLV I and II negative
* No other uncontrolled illness, underlying medical condition, psychiatric illness, or social situation that would preclude study participation
* No ongoing or active infection
* No active autoimmune disease requiring treatment
* No significant traumatic injury within the past 4 weeks
* No serious nonhealing wound, ulcer, or bone fracture
* No other "currently active" malignancy except nonmelanoma skin cancer

  * Not "currently active" if considered by physician as having less than 30% risk of relapse after completion of therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No prior anti-vascular endothelial growth factor therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior hormonal therapy (e.g., luteinizing hormone-releasing hormone [LHRH] agonists or antagonists, antiandrogens, estrogens, megestrol, or PC-SPES) for progressive disease
* Prior hormonal therapy in adjuvant or neoadjuvant setting as primary therapy allowed if at least 3 months since androgen deprivation
* No concurrent systemic steroid therapy (inhaled or topical steroids allowed)

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery, including open biopsy or needle biopsy of liver
* No concurrent major surgery

Other:

* At least 10 days since prior aspirin
* At least 10 days since prior oral or parenteral anticoagulants except to maintain patency of pre-existing permanent indwelling IV catheters
* No concurrent aspirin
* No concurrent oral or parenteral anticoagulants except to maintain patency of pre-existing permanent indwelling IV catheters
* No other concurrent experimental or commercial agents or therapies for prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-12; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Small, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States